CLINICAL TRIAL: NCT02125721
Title: Effect of Increasing Doses of Cystine Binding Thiol Drugs on Cystine Capacity in Patients With Cystinuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-00108; 1U54DK083908 (NIH)
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Cystinuria
Keywords: cystinuria; D-penicillamine (Cuprimine®); tiopronin (Thiola®)
MeSH Terms: conditions — Cystinuria | interventions — Tiopronin; Penicillamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CBTD Patients (Experimental): Part 1: patients will stop taking CBTDs for seven days and perform a 24-hour urine collection on day 7 Part 2: patients will take their usual CBTD, either tiopronin or d-penicillamine, 1g per day for 7 days, taken as 500 mg twice a day Part 3: patients will take a total of 2g of tiopronin or D-penicillamine daily for 7 days Part 4: patients will take a total of 3g/d of tiopronin or D-penicillamine, also for a 7 day period
  Interventions: Drug: Tiopronin 1g per day; Drug: Tiopronin 2g per day; Drug: Tiopronin 3g per day

INTERVENTIONS:
Drug: Tiopronin 1g per day — 500mg PO BID x 7 days
  Other Names: Thiola or tiopronin; d-penicillamine
Drug: Tiopronin 2g per day — 1g PO BID x 7 days
  Other Names: Thiola or tiopronin; d-penicillamine
Drug: Tiopronin 3g per day — 1.5g PO BID x 7 days
  Other Names: Thiola or tiopronin; d-penicillamine

SUMMARY:
The purpose of this study is to evaluate the effect of escalating doses of cystine biding thiol drugs, including tiopronin and d-penicillamine, on the urinary cystine capacity, which is a measure of the amount of cystine in the urine, in patients with cystinuria. The overall goal will be to help guide therapy and ultimately minimize unnecessary side effects caused by larger doses.

DETAILED DESCRIPTION:
Cystinuria is a rare genetic cause of kidney stones that leads to significant morbidity due to the recurrent nature of the disease. As a result, a significant part of treatment is focused on prevention of stone formation. Current methods of prevention include increasing fluid intake, dietary modifications, alkali therapy, and cystine binding thiol drugs (CBTDs), which help increase the solubility of cystine in the urine. At present, the dosing of CBTDs is empiric, and not titrated to a specific measured effect. Our primary objective will be to measure the effect of increasing doses of CBTDs on cystine capacity. The investigators predict that higher dosages of these medications will lead to a more positive urinary cystine capacity, or the ability of urine to take up more cystine (and therefore decreased risk of stone formation). However, the dose at which increasing dosages of the medications cease to provide additional benefit is unknown. The investigators will directly measure the cystine capacity in the urine in response to increasing doses of medications to determine if there is a dose at which the maximum benefit of the drug exists.

This is a cross-over trial of escalating doses. There will be four parts to the study. In the first part, subjects will stop taking CBTDs for 7 days, and perform a 24-hour urine collection on day 7. In part 2, they will take their usual CBTD (either tiopronin or d-penicillamine) 1 gram per day for 7 days. They will perform another 24-hour urine collection on day 7 of this study period. In part 3, they will take their usual CBTD at 2 grams per day for 7 days and in part 4 they will take their CBTD at 3 grams per day for 7 days. Again, they will perform 24-hour urine collections on day 7 of each period. The order in which the parts of the study are performed will be randomized for each subject. The mean cystine capacities in each part of the study will be compared to determine the effect of drug dosage on urinary cystine capacity.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient with a confirmed diagnosis of cystinuria.
* Be already taking a CBTD (either D-penicillamine (Cuprimine®) or tiopronin (Thiola®) as part of your medication regimen.
* Be between 18 and 80 years of age
* Be enrolled in the Cystinuria Registry.

Exclusion Criteria:

* You are not a patient with cystinuria
* You are not already taking a cystine binding thiol drug
* You have renal colic (if you are passing a stone)
* You are scheduled to undergo a urologic procedure
* You are unwilling or unable to provide informed consent in order to be able to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldfarb, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow data was not provided "per sequence". Multiple efforts were made to obtain information, but have not been successful.
Period: Overall Study
Arm/Group | CBTD Patients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CBTD Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Cystine Capacity
Description: We will test for a negative correlation between progressive increases in doses of thiol drugs and cystine capacity
Time Frame: 4 weeks on assigned therapy
Population: Multiple efforts to contact the PI/study team for the relevant data have failed. Therefore, per intervention data are not available to be reported for this assessment.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Increasing Doses of CBTD: Intervention: CBTD 0-3 gm
  CBTD 0-3 gm: Oral CBTD 0-3 gm dose/day for 7 days, dose escalation
Arm/Group | Increasing Doses of CBTD
Number analyzed (Participants) | 7
mg/L | 43.1 (131.2)

ADVERSE EVENTS:
Time Frame: 10 Days
Description: Multiple efforts to contact the PI/study team for the relevant data have failed. Therefore, per intervention data are not available to be reported for this assessment.
Arm/Group | CBTD Patients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT02125721/Prot_SAP_000.pdf